CLINICAL TRIAL: NCT06277297
Title: Exploring the eVolution in prognOstic capabiLity of mUlti-sequence Cardiac magneTIc resOnance in patieNts Affected by Takotsubo Cardiomyopathy
Brief Title: Prognotic Role of CMR in Takotsubo Syndrome
Acronym: EVOLUTION
Status: Recruiting | Type: Observational
Sponsor: University of Cagliari (Other)
Collaborators: Centro Cardiologico Monzino (Other); IRCCS San Raffaele (Other); University of Roma La Sapienza (Other); Fondazione C.N.R./Regione Toscana "G. Monasterio", Pisa, Italy (Other Government); University of Messina (Other); University of Udine (Other); Vannini Hospital Rome (Unknown); A.O.U. Città della Salute e della Scienza - Molinette Hospital (Other); University Hospital, Bonn (Other); University Hospital, Rouen (Other)
Responsible Party: Principal Investigator, Riccardo Cau, Principal investigator, University of Cagliari
Other Study IDs: NP/2022/4583
Record Dates: First submitted 2024-02-09; First posted 2024-02-26 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-03

CONDITIONS: Takotsubo Cardiomyopathy; Machine Learning; Magnetic Resonance Imaging
MeSH Terms: conditions — Takotsubo Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The primary objective of this observational registry is to develop a comprehensive clinical and imaging score (incorporating echocardiography and cardiac magnetic resonance data) that enhances risk stratification for patients with Takotsubo syndrome.

The secondary objectives of this registry are as follows:

Investigate the diagnostic value of cardiac magnetic resonance parameters in predicting in-hospital and long-term outcomes in patients with Takotsubo syndrome.

Compare the proposed risk stratification score for patients with Takotsubo syndrome with previously existing scores.

Investigate the contribution of machine learning models in predicting in-hospital and long-term outcomes compared to standard clinical scores.

The design and rationale of this registry are available at 10.1097/RTI.0000000000000709

DETAILED DESCRIPTION:
The prognosis of Takotsubo syndrome patients remains contentious, necessitating improved risk stratification for better management. While various clinical characteristics and parameters from transthoracic echocardiography have been associated with outcomes, none of the existing predictive scores incorporate cardiac magnetic resonance imaging (CMR) data, despite its ability to noninvasively assess tissue characterization. CMR offers a comprehensive evaluation of functional and structural changes, including an accurate assessment of right ventricular function. While CMR has been extensively studied for diagnostic purposes in Takotsubo syndrome, its role in prognosis is still debated. Emerging technologies like computed tomography show promise in myocardial characterization but lack robust investigation in prognostic roles. The EVOLUTION registry aims to address this gap by incorporating CMR parameters into a risk stratification score alongside clinical and transthoracic echocardiography data, with machine learning models also explored for enhanced outcome prediction. This initiative seeks to provide a more reliable predictive tool for the optimized management of Takotsubo syndrome patients. The main objective of this study is to enhance risk assessment in Takotsubo syndrome patients by incorporating CMR data alongside demographic, clinical, and transthoracic echocardiography parameters. Specifically, the aim is to analyze CMR data and their association with both short-term and long-term patient outcomes. Additionally, the effectiveness of the proposed risk stratification score for Takotsubo syndrome patients will be evaluated in comparison to existing scoring systems. Moreover, all available CMR, transthoracic echocardiography, and clinical variables will be utilized to develop machine learning models for predictive analysis

ELIGIBILITY:
Inclusion Criteria:

* Takotsubo syndrome diagnosis (according to Position Statement of the European Society of Cardiology Heart Failure Association)
* Adult patients ( > 18y old)
* Availability at baseline of clinical variables, standard transthoracic echocardiography, and cardiovascular magnetic resonance acquisition

Exclusion Criteria:

* <18 y old
* Lack of transthoracic echocardiography and cardiovascular magnetic resonance examinations
* Preexisting cardiomyopathies
* Previous myocardial infarction
* Suspected or known prior irreversible myocardial damage
* Valvular heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Takotsubo syndrome patients
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality | 2 years
  cardiovascular death, pulmonary edema, arrhythmias, heart failure, sudden car- diac death, and major adverse cardiac and cerebrovascular events (MACCE) defined as a composite endpoint of death from any cause, myocardial infarction, recurrence of Takotsubo syndrome, transient ischemic attack, and stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cagliari, Cagliari, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cau R, Muscogiuri G, Pisu F, Gatti M, Velthuis B, Loewe C, Cademartiri F, Pontone G, Montisci R, Guglielmo M, Sironi S, Esposito A, Francone M, Dacher N, Peebles C, Bastarrika G, Salgado R, Saba L. Exploring the EVolution in PrognOstic CapabiLity of MUltisequence Cardiac MagneTIc ResOnance in PatieNts Affected by Takotsubo Cardiomyopathy Based on Machine Learning Analysis: Design and Rationale of the EVOLUTION Study. J Thorac Imaging. 2023 Nov 1;38(6):391-398. doi: 10.1097/RTI.0000000000000709. Epub 2023 Apr 4. PMID 37015834